CLINICAL TRIAL: NCT00707707
Title: Phase I/II Randomised, Double- Blind, Multi-centre Study to Assess the Efficacy of AZD2281 When Given in Combination With Paclitaxel in the 1st or 2nd Line Treatment of Patients With Metastatic Triple Negative Breast Cancer.
Brief Title: Phase I/II Study of AZD2281 Given in Combination With Paclitaxel in Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00011
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Metastatic Breast Cancer
Keywords: breast cancer; triple negative; metastatic
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — olaparib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): paclitaxel + AZD2281
  Interventions: Drug: AZD2281; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD2281 — Dose finding study to establish the appropriate dose of AZD2281
  Other Names: Olaparib
Drug: Paclitaxel — Intravenous infusion over 1 hour
  Other Names: Taxol

SUMMARY:
This is the first part of a 2-part study assessing the efficacy of AZD2281 in combination with paclitaxel in 1st or 2nd line treatment of patients with metastatic triple negative breast cancer. This first part (Phase I) is an open-label, intra patient dose finding study to establish the appropriate doses and schedule of paclitaxel and AZD2281 in combination, to be used in the randomized Phase II part. The safety and tolerability of AZD2281 in combination with paclitaxel will be explored. Approximately 10 patients per cohort from 4-5 countries will be enrolled in Phase I.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically or cytologically diagnosed metastatic triple negative breast cancer (Oestrogen, progesterone and HER2 negative adenocarcinoma of the breast)
* Patients must have normal organ and bone marrow function, ECOG performance status of no more than 2
* Formalin fixed, paraffin embedded tumour sample from the primary or recurrent cancer must be available for central testing.

Exclusion Criteria:

* Any chemotherapy, radiotherapy (except for palliative reasons) or investigational product, within 2 weeks from the last dose prior to study entry (or longer period, depending on the agent used)
* Major surgery within 4 weeks of starting the study, and must have recovered from any effects of major surgery
* Patients requiring treatment with the following:certain antibiotic drugs, St.John's Wort, carbamazepine, phenobarbitone, phenytoin, and certain protease inhibitors/ non-nucleoside reverse transcriptase inhibitors used as components of HIV/AIDS treatment,
* Patients with second primary cancer; except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for at least 5 years.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2009-11-09 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events (AEs), physical examination, vital signs including blood pressure (BP), pulse, electrocardiogram (ECG) and laboratory findings including clinical chemistry, hematology, urinalysis | Physical examination/ ECG approximately monthly.Adverse Events, Vital signs, Haematology/ clinical chemistry, Urinalysis weekly throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Dent, MD, Principal Investigator — Sunnybrook Health Sciences Centre, Toronto; Mark Clemons, MD, Principal Investigator — Princess Margaret Hospital, Toronto; Mika Sovak, MD PhD, Study Director — AstraZeneca
Locations (6):
- Australia (3):
  - Research Site, Auchenflower
  - Research Site, Parkville
  - Research Site, Perth
- Research Site, Vienna, Austria
- Research Site, Leuven, Belgium
- Research Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dent RA, Lindeman GJ, Clemons M, Wildiers H, Chan A, McCarthy NJ, Singer CF, Lowe ES, Watkins CL, Carmichael J. Phase I trial of the oral PARP inhibitor olaparib in combination with paclitaxel for first- or second-line treatment of patients with metastatic triple-negative breast cancer. Breast Cancer Res. 2013;15(5):R88. doi: 10.1186/bcr3484. PMID 24063698
- See also: D0810C00011_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1673&filename=D0810C00011.pdf